CLINICAL TRIAL: NCT01730378
Title: Immunogenicity and Safety of GlaxoSmithKline Biologicals' (Pre-) Pandemic Influenza Vaccine Prepandrix™ in Korean Subjects Aged 18 to 60 Years Old
Brief Title: Immunogenicity and Safety of PrepandrixTM in Korean Subjects Aged 18 to 60 Years Old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114695
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2016-05

CONDITIONS: Influenza
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — halofantrine; Lead; fluarix

ARMS (2):
- Prepandrix Group (Experimental): Subjects in this group received 2 doses of Prepandrix™ vaccine at Days 0 and 21. The vaccine was administered intramuscularly in the deltoid region of arm (non-dominant arm at Day 0 and dominant arm at Day 21).
  Interventions: Biological: Prepandrix™
- Fluarix Group (Active Comparator): Subjects in this group received 1 dose of Fluarix™ vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid region of non-dominant arm.
  Interventions: Biological: Fluarix™

INTERVENTIONS:
Biological: Prepandrix™ — 2 doses administered intramuscularly in the deltoid region of arm (non-dominant arm at Day 0 and dominant arm at Day 21).
  Other Names: GlaxoSmithKline [GSK] Biologicals' A/Indonesia/5/2005 (H5N1) (pre-) pandemic influenza adjuvanted vaccine
  Arms: Prepandrix Group
Biological: Fluarix™ — 1 dose administered intramuscularly in the deltoid region of non-dominant arm.
  Other Names: GSK Biologicals' trivalent inactivated influenza split vaccine (Influsplit SSW® 2012/2013)
  Arms: Fluarix Group

SUMMARY:
This study will evaluate the immunogenicity and the safety of PrepandrixTM in Korean subjects. A second group of subjects will receive FluarixTM vaccine as control.

DETAILED DESCRIPTION:
Initially, 124 subjects were planned to be enrolled according to a 1:1 randomisation ratio. However, by mistake, the randomisation application was set up consistent with the vaccine supply ratio (2:1) rather than the treatment group randomization ratio (1:1). Subsequently, the protocol was amended to adjust the sample size and randomisation ratio for the study.

The study will enrol 126 subjects randomised 2:1. 84 subjects will receive Prepandrix™ and 42 subjects will receive Fluarix™.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol. Or subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) can and will comply with the requirements of the protocol.
* Korean male or female subject between, and including, 18 and 60 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject/ from the parent(s)/ Legally Acceptable Representative(s).
* Healthy subjects or free of acute aggravation of the health status as established by medical history and clinical examination before entering into the study.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject has practiced adequate contraception for 30 days prior to vaccination, has a negative pregnancy test on the day of vaccination, and has agreed to continue adequate contraception during the entire treatment period and for two months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Acute disease and/or fever at the time of enrollment.
* Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Diagnosed with cancer, or treatment for cancer, within the past three years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including history of human immunodeficiency virus (HIV) infection.
* Family history of congenital or hereditary immunodeficiency.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without any clinically-apparent bleeding tendency, are eligible.
* History of any neurological disorders or seizures.
* An acute evolving neurological disorder or history of Guillan-Barré syndrome.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Any administration of long-acting immune-modifying drugs within three months before study start, or a planned administration during the study period.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Clinically or virologically diagnosed influenza infection within six months preceding the study start.
* Administration of any vaccines within 30 days before vaccination, or planned administration during the study start.
* Previous vaccination against influenza with any seasonal or pandemic vaccine within six months preceding the administration of the study vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* History of allergy or reactions likely to be exacerbated by any component of the vaccines, including history of a severe adverse reaction to a previous dose of influenza vaccine.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Child in care.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2012-12-05; Primary Completion 2013-12-17 (Actual); Study Completion 2013-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- South Korea (4):
  - GSK Investigational Site, Guro Gu
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul

REFERENCES:
- [Derived] Izurieta P, Kim WJ, Wie SH, Lee J, Lee JS, Drame M, Vaughn DW, Schuind A. Immunogenicity and safety of an AS03-adjuvanted H5N1 pandemic influenza vaccine in Korean adults: a phase IV, randomized, open-label, controlled study. Vaccine. 2015 Jun 4;33(24):2800-7. doi: 10.1016/j.vaccine.2015.04.027. Epub 2015 Apr 21. PMID 25910919

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prepandrix Group | Fluarix Group
Started | 84 | 47
Completed | 83 | 47
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prepandrix Group | Fluarix Group | Total
Number analyzed (Participants) | 84 | 47 | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (10.94) | 40.4 (10.3) | 39.69 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 34 | 95
  Male | 23 | 13 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Serum H5N1 Haemagglutination-inhibition (HI) Antibodies Against Flu A/Indonesia/5/2005 (H5N1) Vaccine Strain in Prepandrix Group.
Description: A seroconverted subjects was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer.
Time Frame: At Day 42
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity included all evaluable subjects for whom data concerning immunogenicity outcome variables were available. This included subjects for whom assay results were available for antibodies against at least 1 study vaccine antigen component after vaccination.
Measure: Number; unit: Subjects
Arm/Group | Prepandrix Group
Number analyzed (Participants) | 81
Subjects | 81

2. Primary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Flu A/Indonesia/5/2005 (H5N1) Vaccine Strain in Prepandrix Group.
Description: MGI was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination (Day 0).
Time Frame: At Day 42
Population: Analysis was performed on the ATP cohort for immunogenicity included all evaluable subjects for whom data concerning immunogenicity outcome variables were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Prepandrix Group
Number analyzed (Participants) | 81
Fold increase | 58.0 [48.7 to 69.1]

3. Primary Outcome: Number of Subjects Who Were Seroprotected for Anti-HI Antibodies Against Flu A/Indonesia/5/2005 (H5N1) Vaccine Strain in Prepandrix Group.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40 that usually is accepted as indicating protection in adults.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Prepandrix Group
Number analyzed (Participants) | 81
Subjects | 81

4. Primary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibody Titers Against Flu A/Indonesia/5/2005 (H5N1) Vaccine Strain in Prepandrix Group.
Description: Antibody titers were expressed as Geometric mean titers (GMTs).
Time Frame: At Day 0 and Day 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Prepandrix Group
Number analyzed (Participants) | 81
Titer
  H5N1, Day 0 | 5.2 [5.0 to 5.3]
  H5N1, Day 42 | 300.1 [254.1 to 354.5]

5. Secondary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibody Titers Against Against Flu A/Indonesia/5/2005 (H5N1) Vaccine Strain in Prepandrix Group.
Description: Antibody titers were expressed as Geometric mean titers (GMTs).
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Prepandrix Group
Number analyzed (Participants) | 81
Titer | 31.8 [26.2 to 38.7]

6. Secondary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against Flu A/Indonesia/5/2005 (H5N1) Vaccine Strain in Prepandrix Group.
Description: as for outcome 3
Time Frame: At Day 0 and Day 21
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Prepandrix Group
Number analyzed (Participants) | 81
Subjects
  H5N1, Day 0 | 0
  H5N1, Day 21 | 37

7. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against Flu A/Indonesia/5/2005 (H5N1) Vaccine Strain in Prepandrix Group.
Description: as for outcome 1
Time Frame: At Day 21
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Prepandrix Group
Number analyzed (Participants) | 81
Subjects | 37

8. Secondary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Flu A/Indonesia/5/2005 (H5N1) Vaccine Strain in Prepandrix Group.
Description: MGI was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination (Day 0).
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Prepandrix Group
Number analyzed (Participants) | 81
Fold increase | 6.2 [5.1 to 7.5]

9. Secondary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibody Titers Against Each of the Three Vaccine Seasonal Influenza Strains in Fluarix Group.
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Victoria/361/2011 (H3N2) and Flu B/Hubei-Wujiagang/158/2009 (Yamagata).
Time Frame: At Days 0 and 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluarix Group
Number analyzed (Participants) | 40
Titer
  H1N1, Day 0 | 18.3 [12.0 to 27.9]
  H1N1, Day 21 | 425.9 [289.9 to 625.7]
  H3N2, Day 0 | 22.0 [14.7 to 33.0]
  H3N2, Day 21 | 149.2 [108.5 to 205.3]
  Yamagata, Day 0 | 60.1 [43.0 to 84.0]
  Yamagata, Day 21 | 367.6 [304.7 to 443.4]

10. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against Each of the Three Vaccine Seasonal Influenza Strains in Fluarix Group.
Description: A seroconverted subjects was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Victoria/361/2011 (H3N2)and Flu B/Hubei-Wujiagang/158/2009 (Yamagata).
Time Frame: At Day 21
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group
Number analyzed (Participants) | 40
Subjects
  H1N1 | 33
  H3N2 | 24
  Yamagata | 26

11. Secondary Outcome: Mean Geometric Increase (MGI) for HI Antibodies Against Each of the Three Vaccine Seasonal Influenza Strains in Fluarix Group.
Description: MGI was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination (Day 0). The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Victoria/361/2011 (H3N2) and Flu B/Hubei-Wujiagang/158/2009 (Yamagata).
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluarix Group
Number analyzed (Participants) | 40
Fold increase
  H1N1 | 23.3 [13.7 to 39.3]
  H3N2 | 6.8 [4.3 to 10.7]
  Yamagata | 6.1 [4.3 to 8.7]

12. Secondary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against Each of the Three Vaccine Seasonal Influenza Strains in Fluarix Group.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40 that usually is accepted as indicating protection in adults. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Victoria/361/2011 (H3N2) and Flu B/Hubei-Wujiagang/158/2009 (Yamagata).
Time Frame: At Day 0 and Day 21
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group
Number analyzed (Participants) | 40
Subjects
  H1N1, Day 0 | 14
  H1N1, Day 21 | 39
  H3N2, Day 0 | 15
  H3N2, Day 21 | 38
  Yamagata, Day 0 | 30
  Yamagata, Day 21 | 40

13. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as significant pain at rest that prevented normal everyday activities as assessed by inability to attend/do work or school. Grade 3 redness and swelling was greater than 100 millimeters (mm) i.e. >100mm.
Time Frame: During the 7-day (Day 0-6) period after each vaccination
Population: Analysis was performed on the Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Prepandrix Group | Fluarix Group
Number analyzed (Participants) | 84 | 47
Subjects
  Any Pain | 80 | 32
  Grade 3 Pain | 8 | 0
  Any Redness | 27 | 6
  Grade 3 Redness | 0 | 0
  Any Swelling | 16 | 2
  Grade 3 Swelling | 0 | 0

14. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were fatigue, headache, joint pain, muscle aches, shivering, increased sweating and fever [axillary temperature above 38.0 degrees Celsius (°C)]. Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity as assessed by inability to attend/do work or school, or requires intervention of a physician/healthcare provider. Grade 3 fever = axillary temperature above 39.0°C
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: Analysis was performed on the Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Prepandrix Group | Fluarix Group
Number analyzed (Participants) | 84 | 47
Subjects
  Any Fatigue | 54 | 14
  Grade 3 Fatigue | 4 | 0
  Related Fatigue | 51 | 13
  Any Headache | 38 | 8
  Grade 3 Headache | 4 | 0
  Related Headache | 37 | 5
  Any Increased Sweating | 28 | 3
  Grade 3 Increased Sweating | 2 | 0
  Related Increased Sweating | 28 | 3
  Any Joint Pain | 30 | 5
  Grade 3 Joint Pain | 5 | 0
  Related Joint Pain | 30 | 5
  Any Muscle Aches | 62 | 13
  Grade 3 Muscle Aches | 6 | 0
  Related Muscle Aches | 61 | 13
  Any Shivering | 32 | 4
  Grade 3 Shivering | 3 | 0
  Related Shivering | 32 | 4
  Any Fever (≥ 38.0°C) | 2 | 0
  Grade 3 Fever (≥ 39.0°C) | 0 | 0
  Related Fever | 2 | 0

15. Secondary Outcome: Number of Subjects Reporting Any Potential Immune Mediated Diseases (pIMDs).
Description: Potential immune-mediated diseases (pIMDs) were defined as a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: During the entire study period (From Day 0 to Day 182)
Population: Analysis was performed on the Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Prepandrix Group | Fluarix Group
Number analyzed (Participants) | 84 | 47
Subjects | 0 | 0

16. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 21 days (Day 0-20) post-vaccination period
Population: Analysis was performed on the Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Prepandrix Group | Fluarix Group
Number analyzed (Participants) | 84 | 47
Subjects | 28 | 9

17. Secondary Outcome: Number of Subjects Reporting Unsolicted AEs
Description: as for outcome 16
Time Frame: During the 84-day (Days 0-83) post vaccination period
Population: Analysis was performed on the Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Prepandrix Group | Fluarix Group
Number analyzed (Participants) | 84 | 47
Subjects | 29 | 12

18. Secondary Outcome: Number of Subjects Any Unsolicited AEs
Description: as for outcome 16
Time Frame: During the 63-day (Days 21-83) post-dose 2 in Prepandrix Group
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Prepandrix Group
Number analyzed (Participants) | 84
Subjects | 16

19. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: A serious adverse event was any untoward medical occurrence that: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (From Day 0 to 182)
Population: Analysis was performed on the Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Prepandrix Group | Fluarix Group
Number analyzed (Participants) | 84 | 47
Subjects
  Any SAEs | 1 | 0
  Related SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 to Day 182; Solicited local and general symptoms: During the 7-day (Days 0-6) post-vaccination period; Unsolicited symptoms: During the 84-day (Day 0-83) post-vaccination period
Arm/Group | Prepandrix Group | Fluarix Group
Serious Adverse Events (participants affected / at risk) | 1/84 | 0/47
Other Adverse Events (participants affected / at risk) | 81/84 | 40/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prepandrix Group (N=84) | Fluarix Group (N=47)
Appendicitis (Infections and infestations) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prepandrix Group (N=84) | Fluarix Group (N=47)
Pain (General disorders) | 80 | 32
Redness (General disorders) | 27 | 6
Swelling (General disorders) | 16 | 2
Fatigue (General disorders) | 54 | 14
Headache (General disorders) | 38 | 8
Increased Sweating (General disorders) | 28 | 3
Joint Pain (General disorders) | 30 | 5
Muscles Aches (General disorders) | 62 | 13
Shivering (General disorders) | 32 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.